CLINICAL TRIAL: NCT03481348
Title: Pharyngeal Electrical Stimulation in Amyotrophic Lateral Sclerosis: A Pilot Study With 20 Patients
Brief Title: Pharyngeal Electrical Stimulation in Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., Prof., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PES-ALS
Record Dates: First submitted 2018-03-08; First posted 2018-03-29 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharyngeal Electrical Stimulation (Experimental): PES for 10 minutes per day on 3 consecutive days in addition to standard therapy (logopedic counselling, advice for nutrition, learning of swallowing techniques)
  Interventions: Device: Pharyngeal Electrical Stimulation
- Control (No Intervention): Standard therapy (logopedic counselling, advice for nutrition, learning of swallowing techniques)

INTERVENTIONS:
Device: Pharyngeal Electrical Stimulation — Pharyngeal Electrical Stimulation is applied at the pharynx via a nasogastral tube for 10 minutes per day on 3 consecutive days.
  Arms: Pharyngeal Electrical Stimulation

SUMMARY:
During the course of ALS most patients develop swallowing deficits. In this pilot study we investigate if dysphagia in ALS can be improved by Pharyngeal Electrical Stimulation (PES). PES is Communauté Européenne (CE-) certificated and has been approved for treatment of neurological, oropharyngeal dysphagia. During PES, electrical stimuli are applied at the pharynx via a nasogastral tube with the aim of triggering reorganization processes in damaged brain structures. There is evidence of a positive effect of PES in Stroke and Multiple Sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* possible, probable or definite ALS according to the revised El Escorial criteria (Brooks et al. 2000)
* age >18 years
* able to understand all information and to give full consent according to good clinical practice (GCP)
* moderate ot severe dysphagia, defined by a mean value (all consistencies) of 4

Exclusion Criteria:

* concurrent participation in another interventional trial
* tracheostomy
* severe psychiatric disorder or clinically manifest dementia
* pulmonal or cardial disorder which constitutes a risk when inserting the tube into the pharynx
* permanent cardiac pacemaker or defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Penetration Aspiration Scale (PAS) Score | day 0 (=before PES), day 4 (=after PES), day 7, day 21, day 90
  Degree of Penetration and Aspiration evaluated by fiberendoscopic evaluation of swallowing (FEES)

SECONDARY OUTCOMES:
Swallowing-Quality of Life Score (SWAL-QOL) | day 0 (=before PES), day 4 (=after PES), day 7, day 21, day 90
  swallowing-specific quality of life questionnaire
Schluckbeeinträchtigungs-Skala (SBS) Score | day 0 (=before PES), day 4 (=after PES), day 7, day 21, day 90
  Clinical scale to evaluate severity of dysphagia
Functional Oral Intake Scale (FOIS) Score | day 0 (=before PES), day 4 (=after PES), day 7, day 21, day 90
  Clinical scale to evaluate the impairment of oral food intake
Dysphagia Severity Rating Scale (DSRS) Score | day 0 (=before PES), day 4 (=after PES), day 7, day 21, day 90
  Clinical scale to evaluate severity of dysphagia
Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALS-FRS-R) | day 0 (=before PES), day 4 (=after PES), day 7, day 21, day 90
  Clinical scale to evaluate the severity of symptoms in ALS
Frequency of Adverse Events | day 0 (=before PES), day 4 (=after PES), day 7, day 21, day 90
  Frequency of Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks BR, Miller RG, Swash M, Munsat TL; World Federation of Neurology Research Group on Motor Neuron Diseases. El Escorial revisited: revised criteria for the diagnosis of amyotrophic lateral sclerosis. Amyotroph Lateral Scler Other Motor Neuron Disord. 2000 Dec;1(5):293-9. doi: 10.1080/146608200300079536. No abstract available. PMID 11464847
- [Derived] Herrmann C, Schradt F, Lindner-Pfleghar B, Schuster J, Ludolph AC, Dorst J. Pharyngeal electrical stimulation in amyotrophic lateral sclerosis: a pilot study. Ther Adv Neurol Disord. 2022 Feb 8;15:17562864211068394. doi: 10.1177/17562864211068394. eCollection 2022. PMID 35154390